CLINICAL TRIAL: NCT04720612
Title: COVID-19 Immunologic Antiviral Therapy With Omalizumab - An Adaptive Phase II Randomized-Controlled Clinical Trial
Brief Title: COVID-19 Immunologic Antiviral Therapy With Omalizumab
Acronym: CIAO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Elena Netchiporouk, Junior Scientist and Assistant Professor of Dermatology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CIAO (2021-7500)
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: Omalizumab; Interferon-alpha; COVID-19; SARS-CoV-2; Coronavirus; Corona virus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omalizumab (Experimental): Participants in this arm will receive the study drug, omalizumab.
  Interventions: Biological: Omalizumab
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Omalizumab — Single subcutaneous dose of 375mg of omalizumab and standard of care.
  Other Names: Xolair
  Arms: Omalizumab
Other: Placebo — Single subcutaneous dose of normal saline in a syringe identical to that of the omalizumab arm and standard of care.
  Arms: Placebo

SUMMARY:
To evaluate if omalizumab is effective in decreasing mortality in severe hospitalized COVID-19 cases.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) has affected over 88 million people, resulting in the death of at least 1.9 million individuals and numbers continue to climb exponentially. Despite these staggering numbers, there are currently very few effective treatments for COVID-19. The immune response to COVID-19 virus appears to follow 2 phases. During the incubation and early disease, interferon (ex. INF-α) signaling and adaptive immunity preclude the disease from progressing. If, and when, this immune response is impaired, the virus may cause pathologic inflammation leading to massive organ dysfunction leading to acute respiratory distress syndrome (ARDS).

Omalizumab is a humanized anti-IgE antibody approved by Health Canada for the treatment of moderate-severe asthma and chronic spontaneous urticaria. Omalizumab has been shown to exhibit antiviral and anti-inflammatory effects in virally exacerbated asthma cases that may be relevant to the treatment of COVID-19.

This is a double blind randomized placebo-controlled trial to evaluate the efficacy of a single dose of omalizumab in reducing all cause mortality at day 29 in severe hospitalized COVID-19 cases. Moreover, time to improvement/hospital discharge, incidence and duration of mechanical ventilation and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Positive RT-PCR assay for SARS-CoV-2;
2. COVID-19 disease requiring hospitalization
3. Dyspnea at rest or during minimal activity (sitting, talking, coughing, swallowing), OR

   * Respiratory rate > 22/min, OR
   * PaO2 < 65mmHg or O2Sat < 90%, OR
   * Infiltrate on chest radiography (CXR) (worsening CXR if baseline abnormal)
4. Age ≥18 years;
5. Ability to provide consent or to provide consent via a substitute decision maker

Patients who are pregnant may also be eligible if consent is provided. Patients who have received one of the SARS-CoV2 vaccines and/or bamlanivimab are eligible to participate in the study

Exclusion Criteria:

1. Known hypersensitivity to Omalizumab or its excipients
2. Inability to give consent themselves or via proxy
3. Patients who received Omalizumab or another anti-IgE molecule in the last 12 months
4. Patients receiving another monoclonal antibody to treat SARS-CoV-2/other indication prior to starting CIAO trial. However, once the study is initiated, if it is judged by the treating team/patient's doctor that patient's health/clinical status may benefit from a monoclonal antibody (e.g. tocilizumab), this will be allowed.
5. Patients who are below the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Death or Mechanical Ventilation | 14 Days
  Outcome reported as the number of patients in each arm that either experience death by any cause or mechanical ventilation.

SECONDARY OUTCOMES:
Time to Clinical Improvement | 28 Days
  Outcome reported as the time to improvement of 2 points on the 8-category ordinal scale. (World Health Organization, 2020)
  8-category ordinal scale: 0- Uninfected, no clinical or virological evidence of infection
  1. Ambulatory, no limitation of activities
  2. Ambulatory, limitation of activities
  3. Hospitalized mild disease, no oxygen therapy
  4. Hospitalized mild disease, oxygen by mask or nasal prongs
  5. Hospitalized severe disease, non invasive ventilation or high-flow oxygen
  6. Hospitalized severe disease, intubation and mechanical ventilation
  7. Hospitalized severe disease, ventilation + additional organ support - pressors, RRT, ECMO
  8. Death
Duration of Mechanical Ventilation | 28 Days
  Outcome reported as duration of mechanical ventilation in each arm.
Duration of Hospitalization | 28 Days
  Outcome reported as the duration of hospitalization of patients in each arm.
Safety in COVID-19 patients | 14 Days
  Outcome reported as the number of adverse events and serious adverse events that occurred in each arm.
Incidence of All-Cause in Hospital Mortality | 28 Days
  Outcome reported as the number of patients in each arm that experience death by any cause while in hospital.

OTHER OUTCOMES:
Percent of viral clearance of Omalizumab as compared to the control arm | Days 0, 2, 7, 14
  Evaluation of the virologic efficacy of omalizumab as compared to the control arm as assessed by the percent of subjects with SARS-CoV-2 detectable in OP/NP sample at days 0, 2, 7, 14.
Spirometry results: Forced Vital Capacity | 6 months
  Evaluation of forced vital capacity, reported in liters, in both omalizumab and control arms at 6 months.
Spirometry results : Forced expiratory volume in one second | 6 months
  Evaluation of forced expiratory volume in one second, reported in liters, in both omalizumab and control arms at 6 months.
Anti-Inflammatory effects of Omalizumab as compared to the control arm | Days 0, 2, 7, 14
  Assessed by measuring cytokine levels, TNF-α, IL-1, IL-6, and IFN-α in picograms per milliliter on days 0, 2, 7, 14.
Anti-fibrotic effects of Omalizumab as compared to the control arm | Days 0, 2, 7, 14
  Assessed by measuring TGF-β level in nanograms per milliliter on days 0, 2, 7, 14.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Netchiporouk, MD, MSc, Principal Investigator — RI-MUHC
Locations (3):
- Canada (3):
  - Niagara Health - St. Catharine's Sites, Niagara, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. WHO R&D Blueprint novel Coronavirus COVID-19 Therapeutic Trial Synopsis. In. Geneva, Switzerland. 2020.
- [Derived] Le M, Khoury L, Lu Y, Prosty C, Cormier M, Cheng MP, Fowler R, Murthy S, Tsang JLY, Ben-Shoshan M, Rahme E, Golchi S, Dendukuri N, Lee TC, Netchiporouk E. COVID-19 Immunologic Antiviral Therapy With Omalizumab (CIAO)-a Randomized Controlled Clinical Trial. Open Forum Infect Dis. 2024 Feb 23;11(4):ofae102. doi: 10.1093/ofid/ofae102. eCollection 2024 Apr. PMID 38560604